CLINICAL TRIAL: NCT06033560
Title: The Effect of Non-invasive Respiratory Support on Outcome and Its Risks in SARS-COV-2-related Hypoxemic Respiratory Failure
Brief Title: The Effect of Non-invasive Respiratory Support on Outcome and Its Risks in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2)-Related Hypoxemic Respiratory Failure
Acronym: NORMO2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof.dr. L.M.A. Heunks, Professor, Erasmus Medical Center
Other Study IDs: RP-D0C3E4
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: COVID-19; Hypoxemic Respiratory Failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Noninvasive Ventilation; Continuous Positive Airway Pressure; Stretchers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Full analysis: All eligible patients.
  Interventions: Device: High flow nasal oxygen (HFNO, more than 15 L/min)
- P/F ratio subgroups: Patients with a P/F ratio split in groups of <=100; 100-150; 150-200
  Interventions: Device: High flow nasal oxygen (HFNO, more than 15 L/min)
- Respiratory rate subgroups: Patients with a respiratory rate split in groups of <=25; >25 breaths/min
  Interventions: Device: High flow nasal oxygen (HFNO, more than 15 L/min)
- Body mass index (BMI) subgroups: Patients with BMI split in groups of <=25; 25-30; 30-35; >35 kg/m^2
  Interventions: Device: High flow nasal oxygen (HFNO, more than 15 L/min)
- Immunocompromised subgroups: Immunocompromised patients due to medication or an underlined condition.
  Interventions: Device: High flow nasal oxygen (HFNO, more than 15 L/min)
- Intensive care unit (ICU) subgroup: Only patients eligible within 24 hours of ICU admission.
  Interventions: Device: High flow nasal oxygen (HFNO, more than 15 L/min)

INTERVENTIONS:
Device: High flow nasal oxygen (HFNO, more than 15 L/min) — Non-invasive respiratory support strategy
  Other Names: Non-invasive ventilation (NIV- Continuous positive airway pressure or bilevel positive airway pressure); Conventional oxygen (COT, between 10 - 15 L/min)

SUMMARY:
Coronavirus disease (COVID-19) can result in severe hypoxemic respiratory failure that ultimately may require invasive mechanical ventilation in the Intensive Care Unit (ICU). Although lifesaving, invasive mechanical ventilation is associated with high mortality, severe discomfort for patient, long-term sequelae, stress to loved-ones and high costs for society. During the ongoing pandemic high number of invasively ventilated COVID-19 patients overwhelmed ICU capacity.

Non-invasive respiratory support, such as high flow nasal oxygen (HFNO) or non-invasive ventilation (NIV) have the potential to reduce the risk for invasive mechanical ventilation and in selected cases ICU admission. However, data from different studies are conflicting and studies performed in COVID-19 patients are of limited quality. Furthermore, identification of early predictors of HFNO/NIV treatment failure may prevent unnecessary delay of initiation of invasive ventilation, which may be associated with adverse clinical outcome. The development and validation of a prediction model, that incorporates readily available clinically data may prove pivotal to fine-tune non-invasive respiratory support.

The overall aim of the NORMO2 project is to investigate the role and risks of HFNO and NIV to improve outcome in hospitalized hypoxemic COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Sars-Cov-2 infection
* hospital admission (emergency department, inpatient or ICU)
* hypoxemic respiratory failure, defined as P/F ratio below or including 200

Exclusion Criteria:

* hypercapnia (PCO2 > 45 mmHG in combination with acidemia (pH < 7.35))
* pregnancy
* do not resuscitate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 hospital sites across the United States
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring invasive mechanical ventilation | 30 days

SECONDARY OUTCOMES:
Mortality at day 30 | 30 days
ICU-free days | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data is accessible through the National COVID Cohort Collaborative website all relevant code for this project will be made available upon completion.